CLINICAL TRIAL: NCT00127075
Title: POPART'MUS: Prevention of Post Partum Relapses With Progestin and Estradiol in Multiple Sclerosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2004.363
Record Dates: First submitted 2005-08-04; First posted 2005-08-05 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis. Relapses. Post partum. Pregnancy. Delivery. Hormones. Progesterone. Estradiol. Clinical trial. Prevention.
MeSH Terms: conditions — Multiple Sclerosis | interventions — nomegestrol acetate; Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NOMA + estradiol (Experimental): Oral NOMA (LUTENYL® 10 mg/day) combined with transdermal Estradiol (DERMESTRIL SEPTEM® 75 mcg, once a week),
  Interventions: Drug: nomegestrol acetate; Drug: estradiol
- placebo (Placebo Comparator): Matching placebo treatments
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: nomegestrol acetate — 10 mg/day
  Arms: NOMA + estradiol
Drug: estradiol — 75 mcg, once a week
  Arms: NOMA + estradiol
Drug: placebo — matching placebo treatments
  Arms: placebo

SUMMARY:
Multiple sclerosis (MS) affects 1 in 1000 people in western countries, mainly women in their childbearing years. It is an autoimmune disease of the central nervous system (CNS), which results in a chronic focal inflammatory response with subsequent demyelination and axonal loss. Recent prospective studies reported a significant decline by two-thirds in the rate of relapses during the third trimester of pregnancy and a significant increase by two-thirds during the first three months post-partum by comparison to the relapse rate observed during the year prior to the pregnancy (Confavreux et al., 1998). These dramatic changes in the relapse rate occur at a time when the impregnation of many substances (among which, sexual steroids) is at its highest, before a dramatic decline to the pre-pregnancy levels, immediately following delivery.

It may be hypothesized that sexual steroids could exert beneficial effects through a modulation of the immune state with a lowering of the pro-inflammatory lymphocyte responses of the Th1 type and an enhancement of the anti-inflammatory responses of the Th2 type. They may also play a direct role in the remyelination of central nervous system lesions, as they do in the peripheral nervous system. The POPART'MUS study is a European, multicentre, randomized, placebo-controlled and double-blind clinical trial, which aims to prevent MS relapses related to the post-partum condition, by administering high doses of progestin (nomegestrol acetate), in combination with endometrial protective doses of estradiol. Treatment will be given immediately after delivery and continuously during the first three months post-partum. Assuming the results of the trial to be positive, this new treatment could be considered in the relapsing-remitting phase of the disease in women afar from pregnancy and post-partum.

ELIGIBILITY:
Inclusion Criteria:

* MS according to MacDonald criteria (including clinically isolated syndromes fulfilling magnetic resonance imaging [MRI] criteria for MS diagnosis)
* Relapsing-remitting or secondary progressive MS
* Expanded disability status scale (EDSS) ≤ 6.0
* Pregnancy ≤ 36 weeks of amenorrhea

Exclusion Criteria:

* Age < 18 years
* Clinical isolated syndrome not fulfilling MacDonald criteria for MS
* Primary progressive MS
* Possible MS or no MS according to MacDonald criteria
* Ongoing or previous myocardial infarction, stroke or venous thromboembolism
* Ongoing or previous breast cancer, or cancer of the uterus
* Severe liver disorder
* Undiagnosed genital bleeding
* Hypersensitivity to one of the study treatments
* Desire for lactation
* Desire for an MS disease-modifying treatment in the 24 weeks after delivery
* Women participating in another trial with a drug
* Refusal of non-hormonal contraception in the 12 weeks following delivery
* Consent form not signed

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2005-06; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
To compare the rate of relapses during the first 12 weeks after delivery, between the treated and placebo groups | 12 weeks

SECONDARY OUTCOMES:
Percentage of patients who remain relapse-free during the 12-week period after delivery | 12 weeks
Rate of relapses, percentage of patients who remain relapse-free during the 24-week period after delivery | 24 weeks
Rate of relapses, percentage of patients who remain relapse-free during the 12- to 24-week period after delivery | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christian Confavreux, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Pierre Wertheimer, Bron, France

REFERENCES:
- [Background] Confavreux C, Hutchinson M, Hours MM, Cortinovis-Tourniaire P, Moreau T. Rate of pregnancy-related relapse in multiple sclerosis. Pregnancy in Multiple Sclerosis Group. N Engl J Med. 1998 Jul 30;339(5):285-91. doi: 10.1056/NEJM199807303390501. PMID 9682040
- [Background] Confavreux C, Hutchinson M, Hours M, Cortinovis-Tourniaire P, Grimaud J, Moreau T. [Multiple sclerosis and pregnancy: clinical issues]. Rev Neurol (Paris). 1999 Mar;155(3):186-91. French. PMID 10339787
- [Background] Vukusic S, Hutchinson M, Hours M, Moreau T, Cortinovis-Tourniaire P, Adeleine P, Confavreux C; Pregnancy In Multiple Sclerosis Group. Pregnancy and multiple sclerosis (the PRIMS study): clinical predictors of post-partum relapse. Brain. 2004 Jun;127(Pt 6):1353-60. doi: 10.1093/brain/awh152. Epub 2004 May 6. PMID 15130950
- [Derived] Vukusic S, Ionescu I, El-Etr M, Schumacher M, Baulieu EE, Cornu C, Confavreux C; Prevention of Post-Partum Relapses with Progestin and Estradiol in Multiple Sclerosis Study Group. The Prevention of Post-Partum Relapses with Progestin and Estradiol in Multiple Sclerosis (POPART'MUS) trial: rationale, objectives and state of advancement. J Neurol Sci. 2009 Nov 15;286(1-2):114-8. doi: 10.1016/j.jns.2009.08.056. Epub 2009 Sep 15. PMID 19758607
- See also: European database for multiple sclerosis — http://www.edmus.org